CLINICAL TRIAL: NCT02603861
Title: An Evaluation of the Impact of Single Doses of LY3154207 on Sleep Latency in Sleep-Deprived Healthy Subjects
Brief Title: A Study of LY3154207 on Sleep in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 15511; I7S-EW-HBEB (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
MeSH Terms: interventions — LY3154207; Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo matching LY3154207 administered once orally in one of four periods.
  Interventions: Drug: Placebo
- LY3154207 - Dose 1 (Experimental): LY3154207 administered orally in no more than one of the four periods.
  Interventions: Drug: LY3154207
- LY3154207 - Dose 2 (Experimental): LY3154207 administered orally in no more than one of the four periods.
  Interventions: Drug: LY3154207
- LY3154207 - Dose 3 (Experimental): LY3154207 administered orally in no more than one of the four periods.
  Interventions: Drug: LY3154207
- Modafinil (Active Comparator): 200 mg modafinil administered orally in no more than one of the four periods.
  Interventions: Drug: Modafinil

INTERVENTIONS:
Drug: LY3154207 — LY3154207 administered orally.
  Arms: LY3154207 - Dose 1; LY3154207 - Dose 2; LY3154207 - Dose 3
Drug: Placebo — Placebo administered orally.
  Arms: Placebo
Drug: Modafinil — Modafinil administered orally.
  Arms: Modafinil

SUMMARY:
This study will evaluate the effect of single doses of LY3154207 on the amount of time it takes for healthy sleep-deprived men to fall asleep. The study will also estimate how much LY3154207 gets into the blood stream and how long it takes the body to remove it. Information about any side effects that occur will be collected. Each participant will complete four study periods, which will last a total of about 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males 18 years of age or older who have given consent and are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have a regular sleep pattern with routine time spent in bed between 6.5 hours and 9 hours each night

Exclusion Criteria:

* Are shift workers who shifted work within 14 days prior to screening or plan to during the study
* Have a known sleep disorder or history of a sleep disorder
* Have traveled 2 time zones or more within 7 days prior to screening or plan to during the study
* Regularly take naps during the day
* Are hearing impaired

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Time to Sleep Onset | Day 1: 2 hours post dose through 8 hours post dose in each period.

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of LY3154207 | Day 1: 1 hour post dose through 24 hours post dose in each period.
Area Under the Concentration Versus Time Curve (AUC) of LY3154207 | Day 1: 1 hour post dose through 24 hours post dose in each period.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Parexel Early Phase Unit at Glendale, Glendale, California, United States